CLINICAL TRIAL: NCT04568772
Title: A Randomized, Open-label, Three-period Crossover Clinical Trial to Evaluate the Influence of Tegoprazan on the Pharmacokinetics of Proguanil in Healthy Volunteers
Brief Title: Study to Evaluate the Influence of Tegoprazan on the Pharmacokinetics of Proguanil in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, SeungHwan Lee, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Tegoprazan_CYP2C19_DDI
Record Dates: First submitted 2020-09-15; First posted 2020-09-29 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Atovaquone; Proguanil; atovaquone, proguanil drug combination; tegoprazan; Esomeprazole; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Atovaquone/Proguanil 250/100 mg (Active Comparator): A single oral administration of atovaquone/proguanil 250/100 mg
  Interventions: Drug: Atovaquone / Proguanil 250/100 mg
- Tegoprazan 50 mg + Atovaquone/Proguanil 250/100 mg (Experimental): Oral administration of tegoprazan 50 mg once daily for 6 days and then co-administration of tegoprazan 50 mg and atovaquone/proguanil 250/100 mg at 7 day
  Interventions: Drug: Atovaquone / Proguanil 250/100 mg; Drug: Tegoprazan 50 mg
- Esomeprazole 40 mg + Atovaquone/Proguanil 250/100 mg (Experimental): Oral administration of esomeprazole 40 mg once daily for 6 days and then co-administration of esomeprazole 40 mg and atovaquone/proguanil 250/100 mg at 7 day
  Interventions: Drug: Atovaquone / Proguanil 250/100 mg; Drug: Esomeprazole 40 mg
- Vonoprazan 20 mg + Atovaquone/Proguanil 250/100 mg (Experimental): Oral administration of vonoprazan 20 mg once daily for 6 days and then co-administration of vonoprazan 20 mg and atovaquone/proguanil 250/100 mg at 7 day
  Interventions: Drug: Atovaquone / Proguanil 250/100 mg; Drug: Vonoprazan 20 mg

INTERVENTIONS:
Drug: Atovaquone / Proguanil 250/100 mg — Atovaquone / Proguanil 250/100 mg tablet
  Other Names: Malarone
Drug: Tegoprazan 50 mg — Tegoprazan 50 mg tablet
  Other Names: K-cab
  Arms: Tegoprazan 50 mg + Atovaquone/Proguanil 250/100 mg
Drug: Esomeprazole 40 mg — Esomeprazole 40 mg tablet
  Other Names: Nexium
  Arms: Esomeprazole 40 mg + Atovaquone/Proguanil 250/100 mg
Drug: Vonoprazan 20 mg — Vonoprazan 20 mg tablet
  Other Names: Takecab
  Arms: Vonoprazan 20 mg + Atovaquone/Proguanil 250/100 mg

SUMMARY:
The aim of this study is to evaluate the influence of tegoprazan on the pharmacokinetics of proguanil in healthy volunteers.

DETAILED DESCRIPTION:
Evaluation criteria

* Pharmacokinetic assessment with plasma concentrations of proguanil and cycloguanil
* Safety assessments with adverse event monitoring including subjective/objective symptoms, physical examination, vital signs, electrocardiogram, and laboratory tests

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged ≥ 19 years and ≤ 50 years at the time of screening
* Body weight of ≥ 55.0 kg and ≤ 90.0 kg, with body mass index (BMI) of ≥ 19.0 kg/m2 and ≤ 30.0 kg/m2 at the time of screening
* Extensive metabolizer (*1/*1) by CYP2C19 genotyping
* A subject without any congenital or chronic disease, and has no medical examination result as pathological symptoms or signs
* A subject who listened to sufficient explanation and fully understood this study, and voluntarily decided to participate and agreed in writing to comply with the precautions
* A subject determined eligible for this study by investigator based physical examination, clinical laboratory tests, interview, etc.

Exclusion Criteria:

* A subject with clinically significant hepatobiliary (severe hepatic impairment, etc.), renal (severe renal impairment, etc.), neurologic, immunologic, respiratory, gastrointestinal, endocrine, blood•oncology, cardiovascular (heart failure, Torsades de pointes, etc.), urinary, or, psychical diseases (except for simple dental past history such as tartar, impacted tooth, or wisdom tooth) or a history
* A subject who has hypersensitivity to the investigational products, drugs containing the same class, or other drugs (penicillin and antibiotics, etc.), or a history of clinically significant hypersensitivity
* A subject with a history of gastrointestinal disorders (gastrointestinal ulcer, gastritis, gastrospasm, gastroesophageal reflux disease, Crohn's disease, etc.) or surgery (except for simple appendectomy and herniotomy) that may affect the safety and pharmacokinetics of the investigational products
* A subject with the following results in the screening test:
* Blood AST (GOT), ALT (GPT): > Normal range upper × 1.5
* Creatinine clearance calculated by MDRD equation: < 80mL/min
* QTc interval: > 450 ms
* Fasting serum glucose: > 126 mg/dL
* Positive serological test (syphilis test, hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test)
* A subject with systolic blood pressure < 90 mmHg or > 150 mmHg, or diastolic blood pressure < 50 mmHg or > 100 mmHg when vital signs are measured in sitting position after resting for at least 3 minutes
* A subject with a history of or positive urine screening for drug abuse
* A subject who administered any prescription drugs or herbal medicine within 2 weeks prior to the expected date of the first dose, or any over-the-counter drug (OTC drug, health functional food or vitamin within 1 week prior to the expected date of the first dose (However, can participate in the study if otherwise decided eligible by the investigator), or is expected to administer it
* A subject who administered drugs that induce or inhibit the drug metabolizing enzymes, such as barbitals, within 1 week prior to the expected date of the first dose
* A subject who participated in other clinical trial or bioequivalence study within 6 months prior to the expected date of the first dose
* A subject who donated whole blood within 2 months or the component blood within 1 month prior to the expected date of the first dose, or received blood transfusion within 1 month prior to the expected date of the first dose
* A subject with persistent alcohol intake (> 21 units/week, 1 unit = 10 g of pure alcohol), or inability to abstain from drinking from 3 days before the expected date of the first dose until the last discharge
* A subject who is a currently smoker (But, can be eligible if he or she quitted smoking 3 months ago), or is not able to cease smoking from 3 months before the expected date of the first dose until the last discharge
* A subject with inability to refrain from grapefruit-containing food from 3 days before the expected date of the first dose until the last discharge
* A subject with excessive caffeine intake (> 5 units/day), or inability to refrain from caffeine or caffeine-containing food from 3 days before the expected date of the first dose until the last discharge
* A subject with inability to use a medically acceptable double contraception or contraception throughout the study and for at least 4 weeks after the last dose, and with inability to agree to donate sperm until the period

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
AUClast of proguanil, cycloguanil | Pre-dose(0 hour) and up to 48 hours in each period
  Systemic exposure of proguanil and cycloguanil

SECONDARY OUTCOMES:
Cmax of proguanil | Pre-dose(0 hour) and up to 48 hours in each period
  Secondary pharmacokinetic parameters of proguanil
AUCinf of proguanil | Pre-dose(0 hour) and up to 48 hours in each period
  Secondary pharmacokinetic parameters of proguanil
Tmax of proguanil | Pre-dose(0 hour) and up to 48 hours in each period
  Secondary pharmacokinetic parameters of proguanil
t1/2 of proguanil | Pre-dose(0 hour) and up to 48 hours in each period
  Secondary pharmacokinetic parameters of proguanil
CL/F of proguanil | Pre-dose(0 hour) and up to 48 hours in each period
  Secondary pharmacokinetic parameters of proguanil
Vz/F of proguanil | Pre-dose(0 hour) and up to 48 hours in each period
  Secondary pharmacokinetic parameters of proguanil
fe of proguanil | Pre-dose(0 hour) and up to 48 hours in each period
  Secondary pharmacokinetic parameters of proguanil
CLR of proguanil | Pre-dose(0 hour) and up to 48 hours in each period
  Secondary pharmacokinetic parameters of proguanil

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang E, Ji SC, Jang IJ, Lee S. Evaluation of CYP2C19-Mediated Pharmacokinetic Drug Interaction of Tegoprazan, Compared with Vonoprazan or Esomeprazole. Clin Pharmacokinet. 2023 Apr;62(4):599-608. doi: 10.1007/s40262-023-01228-4. Epub 2023 Mar 10. PMID 36897544